CLINICAL TRIAL: NCT00243919
Title: Locomotor Experience Applied Post Stroke (LEAPS) Trial
Brief Title: Locomotor Experience Applied Post Stroke Trial
Acronym: LEAPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006846; R01NS050506 (NIH)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2012-12

CONDITIONS: Stroke
Keywords: stroke; locomotor; exercise; walking; training program; body weight support training; physical therapy
MeSH Terms: conditions — Stroke; Motor Activity

ARMS (3):
- Early Locomotor Training Program (Active Comparator): body weight supported training program with treadmill
  Interventions: Behavioral: Early locomotor training program
- Late Locomotor Training Program (Active Comparator): body weight supported training program with treadmill
  Interventions: Behavioral: Late locomotor training program
- Early Home Exercise Program (Active Comparator): a non-specific low intensity exercise program
  Interventions: Behavioral: Home Exercise Program

INTERVENTIONS:
Behavioral: Early locomotor training program — The early locomotor training program is an out-patient program of locomotor training for 36 sessions, 3 times per week, using a body weight support system and stepping on a treadmill and overground training beginning at 2 months post-stroke.
  Other Names: E-LTP; LTP-early
  Arms: Early Locomotor Training Program
Behavioral: Late locomotor training program — The late locomotor training program is an out-patient program of locomotor training for 36 sessions, 3 times per week, using a body weight support system and stepping on a treadmill and overground training beginning at 6 months post-stroke.
  Other Names: L-LTP; LTP-late
  Arms: Late Locomotor Training Program
Behavioral: Home Exercise Program — Participants in the early home exercise group will receive a non-specific low intensity exercise program beginning at 2 months post stroke.
  Other Names: HEP
  Arms: Early Home Exercise Program

SUMMARY:
The purpose of this study is to compare two different treatments to improve walking after stroke (or post-stroke).

DETAILED DESCRIPTION:
The impact of stroke on walking is significant, with only 37 percent of stroke survivors able to walk after the first week after stroke (or post-stroke). Even among those who achieve independent ambulation, significant residual deficits persist in balance and gait speed with a 73 percent incidence of falls among individuals with mild to moderate impairment 6 months post-stroke. Body weight supported treadmill training is one therapeutic method for locomotor training that is rapidly being adopted into physical rehabilitation to improve walking after stroke.

The purpose of this multi-center, randomized controlled study is to compare two different treatments to improve walking after stroke. The two treatments are: 1) a training program that includes use of a body weight support system and a treadmill to practice walking and 2) a physical therapist monitored exercise program to work on general conditioning and strengthening in the patient's home. In addition, investigators will determine the best time to provide training after a stroke and if the training is beneficial for mild, moderate, or severe cases of stroke.

Four hundred subjects will be recruited from five facilities in Florida and California. Screening and subject recruitment will take place within 45 days post-stroke. All stroke patients will be screened to determine eligibility for the study. Eligible subjects will be followed for 2 months post-stroke. At that time, those who are eligible for enrollment and who consent to participate will undergo an exercise tolerance test and baseline assessment. Following this evaluation, participants will be randomized into one of three groups, according to the severity of their locomotor impairment: early locomotor, late locomotor, or early home exercise.

The early locomotor training group will begin the locomotor training program immediately (2 months post stroke). The locomotor training program is an out-patient program of locomotor training for 36 sessions, 3 times per week, using a body weight support system and stepping on a treadmill. The late locomotor training group will begin locomotor training at 6 months post-stroke. Participants in the early home exercise group will receive a non-specific low intensity exercise program beginning immediately (2 months post stroke).

ELIGIBILITY:
Inclusion Criteria:

* Age >/=18
* Stroke within 45-days
* Residual paresis in the lower extremity (fugl-meyer le motor score < 34)
* Ability to sit unsupported for 30 seconds
* Ability to walk at least 10 feet with maximum 1 person assist
* Ability to follow a three step command
* Provision of informed consent
* A self-selected 10 meter gait speed less than 0.8 m/s at the 2-month post-stroke assessment
* Successful completion of an exercise tolerance test

Exclusion Criteria:

* Lived in nursing home prior to stroke
* Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking less than 200 meters
* Serious cardiac conditions (history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living). Anyone meeting New York Heart Association criteria for Class 3 or Class 4 heart disease will be excluded
* History of serious chronic obstructive pulmonary disease or oxygen dependence
* Severe weight bearing pain
* Preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia, or previous stroke with residual neurological deficits
* History of major head trauma
* Lower extremity amputation
* Non-healing ulcers on the lower extremity
* Renal dialysis or end stage liver disease
* Legal blindness or severe visual impairment
* A history of significant psychiatric illness defined by diagnosis of bipolar affective disorder, psychosis, schizophrenia or medication refractory depression
* Life expectancy less than one year
* Severe arthritis or orthopedic problems that limit passive ranges of motion of lower extremity (knee flexion contracture of -10°, knee flexion Range of Motion (ROM) < 90°, hip flexion contracture > 25°, and ankle plantar flexion contracture > 15°
* History of sustained alcoholism or drug abuse in the last six months
* Major post-stroke depression as measured by the Patient Health Questionnaire(PHQ-9 >/= 10) that is not medically managed with antidepressant medication and/or psychotherapy
* History of pulmonary embolism within 6 months
* Uncontrollable diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Severe hypertension with systolic greater than 200 mmHg and diastolic greater than 110 mmHg at rest,
* Previous or current enrollment in a clinical trial to enhance stroke motor recovery
* Lives more than 50 miles from the training sites
* Unable to travel 3 times per week for outpatient training programs
* Intracranial hemorrhage related to aneurysmal rupture or an arteriovenous malformation (hemorrhagic infarctions will not be excluded)

Inclusion and exclusion criteria will be determined by a chart review, depression screen and subject interview by study physician or study coordinator. After initial chart and subject interview, each subject's treating physician will be asked to review inclusion and exclusion criteria and provide a letter supporting inclusion in the study. All subjects who meet selection criteria must successfully complete an exercise tolerance test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2006-04; Primary Completion 2010-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela W. Duncan, PhD, PT, FAPTA, FAHA, Principal Investigator — Professor and Bette Busch Maniscalco, Doctor of Physical Therapy Division, Research Fellow, Department of Community and Family Medicine, Duke Center for Clinical Health Policy Research; Katherine J. Sullivan, Ph.D., PT, Principal Investigator — Co-Principal Investigator, Division of Biokinesiology and Physical Therapy, University of Southern California, Los Angeles, California; Andrea L. Behrman, Ph.D., PT, Principal Investigator — Co-Principal Investigator, Department of Physical Therapy, Brooks Center for Rehabilitation Studies, University of Florida, and Department of Veteran Affairs Brain Rehabilitation Research Center, Gainesville, Florida; Stanley P. Azen, Ph.D.,, Study Director — Director Data Management Core, Biostatistics Division, Department of Preventive Medicine, University of Southern California, Los Angeles, California; Samuel S. Wu, Ph.D., Study Director — Lead Biostatistician - Investigator, Department of Epidemiology and Health Policy Research, University of Florida; Bruce H. Dobkin, MD, Study Director — Investigator, Department of Neurology, University of California, Los Angeles, California; Stephen E. Nadeau, MD, Study Director — Investigator, Geriatric Research, Education and Clinical Center and the Brain Rehabilitation Research Center, Gainesville VA Medical Center, and the Department of Neurology, University of Florida College of Medicine, Gainesville, Fl
Locations (8):
- United States (8):
  - Centinela Freeman Memorial Hospital, Inglewood, California
  - Long Beach Memorial Hospital, Long Beach, California
  - University of Southern California - PT Associates, Los Angeles, California
  - Sharp Memorial Rehabilitation Center, San Diego, California
  - University of Florida, Gainesville, Florida
  - Brooks Rehabilitation Hospital, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Duke University (Administrative Coordinating Center), Durham, North Carolina

REFERENCES:
- [Derived] Seamon BA, Kautz SA, Velozo CA. Measurement Precision and Efficiency of Computerized Adaptive Testing for the Activities-specific Balance Confidence Scale in People With Stroke. Phys Ther. 2021 Apr 4;101(4):pzab020. doi: 10.1093/ptj/pzab020. PMID 33481989
- [Derived] Nadeau SE, Dobkin B, Wu SS, Pei Q, Duncan PW; LEAPS Investigative Team. The Effects of Stroke Type, Locus, and Extent on Long-Term Outcome of Gait Rehabilitation: The LEAPS Experience. Neurorehabil Neural Repair. 2016 Aug;30(7):615-25. doi: 10.1177/1545968315613851. Epub 2015 Oct 23. PMID 26498434
- [Derived] Nadeau SE, Wu SS, Dobkin BH, Azen SP, Rose DK, Tilson JK, Cen SY, Duncan PW; LEAPS Investigative Team. Effects of task-specific and impairment-based training compared with usual care on functional walking ability after inpatient stroke rehabilitation: LEAPS Trial. Neurorehabil Neural Repair. 2013 May;27(4):370-80. doi: 10.1177/1545968313481284. Epub 2013 Mar 15. PMID 23504552
- [Derived] Tilson JK, Wu SS, Cen SY, Feng Q, Rose DR, Behrman AL, Azen SP, Duncan PW. Characterizing and identifying risk for falls in the LEAPS study: a randomized clinical trial of interventions to improve walking poststroke. Stroke. 2012 Feb;43(2):446-52. doi: 10.1161/STROKEAHA.111.636258. Epub 2012 Jan 12. PMID 22246687
- [Derived] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK, Cen S, Hayden SK; LEAPS Investigative Team. Body-weight-supported treadmill rehabilitation after stroke. N Engl J Med. 2011 May 26;364(21):2026-36. doi: 10.1056/NEJMoa1010790. PMID 21612471
- [Derived] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 inpatient rehabilitation centers in California and Florida from April 2006 through June 2009.
Pre-assignment Details: Participants admitted for inpatient rehabilitation were screened by chart review. Eligible participants with first-time stroke received a comprehensive medical record review and physical and cognitive screening. At 2-months, those who maintained eligibility and successfully completed an exercise tolerance test were enrolled.
Groups:
- Early Locomotor Training Program: Stepping on a treadmill with partial body weight support and manual assistance as needed for 20-30 minutes at 2.0 mph, followed by a progressive overground walking program for 20 minutes delivered at 2 months post-stroke.
- Late Locomotor Training Program: Stepping on a treadmill with partial body weight support and manual assistance as needed for 20-30 minutes at 2.0 mph, followed by a progressive overground walking program for 20 minutes delivered at 6 months post-stroke.
- Home Exercise Program: Home Exercise Program (HEP) was designed as an active control. The exercise program was progressed by a study physical therapist in the home to enhance flexibility, joint range of motion, upper- and lower-extremity strength, coordination and static and dynamic balance. Subjects were encouraged to walk daily. The home exercise program was delivered at 2 months post-stroke.
Period: Overall Study
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Started | 139 | 143 | 126
Completed | 122 | 125 | 115
Not Completed | 17 | 18 | 11
Not completed — Death | 3 | 4 | 6
Not completed — Withdrawal by Subject | 6 | 6 | 2
Not completed — Lost to Follow-up | 6 | 7 | 3
Not completed — Administrative Error | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Home Exercise Program: HEP was designed as an active control. The exercise program was progressed by a study physical therapist in the home to enhance flexibility, joint range of motion, upper- and lower-extremity strength, coordination and static and dynamic balance. Subjects were encouraged to walk daily. The home exercise program was delivered at 2 months post-stroke.
- Total: Total of all reporting groups
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program | Total
Number analyzed (Participants) | 139 | 143 | 126 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.3) | 63.3 (12.5) | 62.6 (13.3) | 62.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 69 | 61 | 184
  Male | 85 | 74 | 65 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 15 | 22 | 63
  Not Hispanic or Latino | 113 | 128 | 104 | 345
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 5
  Asian | 19 | 20 | 15 | 54
  Native Hawaiian or Other Pacific Islander | 4 | 9 | 6 | 19
  Black or African American | 32 | 34 | 24 | 90
  White | 81 | 77 | 78 | 236
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Time since stroke to randomization - days [Mean (Standard Deviation); unit: days] | 64.1 (8.3) | 64.18 (9.0) | 62.9 (8.0) | 63.8 (8.5)
Side of involvement [Number; unit: participants]
  Left Hemiparesis | 63 | 58 | 61 | 182
  Right Hemiparesis | 76 | 85 | 65 | 226
Stroke Type [Number; unit: participants] — Based on CT/MRI overread by study neurologists.
  participants
    Large Vessel | 55 | 60 | 47 | 162
    Lacune | 40 | 45 | 43 | 128
    Hemorrhage | 27 | 22 | 21 | 70
    Undefined | 17 | 16 | 15 | 48
Modified Rankin Scale [Number; unit: participants] — Global measure of stroke disability
  participants
    Rankin 0 - 1 (no significant disability) | 0 | 2 | 0 | 2
    Rankin 2 (slight disability) | 12 | 21 | 21 | 54
    Rankin 3 (moderate disability) | 66 | 57 | 49 | 172
    Rankin 4 (moderately severe disability) | 61 | 63 | 56 | 180
Comorbidities [Number; unit: participants]
  Cardiovascular | 36 | 36 | 37 | 109
  Hypertension | 116 | 111 | 104 | 331
  Peripheral vascular disease | 12 | 12 | 13 | 37
  Chronic Obstructive Pulmonary Disease (COPD) | 5 | 14 | 7 | 26
  Arthritis/other musculoskeletal | 47 | 52 | 47 | 146
  Diabetes | 47 | 51 | 43 | 141
  Depression (Personal Health Questionnaire-9 >= 10) | 20 | 28 | 19 | 67
Mini Mental Status Exam [Mean (Standard Deviation); unit: scores on a scale] — Higher Score is Better;Range = 0-30
  scores on a scale | 26.0 (3.2) | 26.2 (3.7) | 26.0 (3.6) | 26.1 (3.5)
Walking Speed (m/sec) [Number; unit: participants] — Comfortable walking speed assessed by 10 meter walk.
  participants
    Severe Disability (<0.4 m/sec) | 75 | 77 | 66 | 218
    Moderate Disability (0.4 - 0.8 m/sec) | 64 | 66 | 60 | 190
Comfortable walking speed (m/sec) [Mean (Standard Deviation); unit: m/sec] — Assessed with 10 meter walk test.
  m/sec | 0.36 (0.22) | 0.38 (0.23) | 0.39 (0.22) | 0.38 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Successfully Improved Functional Level of Walking at 1 Year Post-stroke
Description: Success: walking greater than 0.4 m/sec if baseline was less than 0.4; walking greater than 0.8 m/sec if baseline was 0.4m/sec or greater but less than 0.8 m/sec as measured during 10 meter walk.
Time Frame: 12 months post-stroke
Population: Intention to treat analysis. Missing data were imputed using the LOCF method.
Measure: Number; unit: percent of participants
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
percent of participants | 50.4 | 53.8 | 51.6
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Home Exercise Program; Logistic regression was used to compare the proportion of participants who improved functional level of walking between Early-LTP and HEP adjusting for pre-specified covariates (severity of impairment, clinical site, age, stroke type, side of hemiparesis and depression). Assuming that 30% of HEP participants would improve functional level of walking, we derived a sample size of 400 to detect a clinically relevant 20% effect size with 85% power, adjusting for an loss-to-follow-up rate of 15%; Test type: Superiority or Other; p = 0.481, Regression, Logistic — The trial tested the superiority of LTP delivered early or late, compared to HEP, using a two-sided significance level of 0.05. The study-wide error rate was controlled by applying the Hochberg step-up procedure to the two primary comparisons; Odds Ratio (OR) = 0.831, 95% CI 2-sided [0.497 to 1.391]
Statistical Analysis 2: Comparison: Late Locomotor Training Program vs Home Exercise Program; Logistic regression was used to compare the proportion of participants who improved functional level of walking between Late-LTP and HEP adjusting for pre-specified covariates (severity of impairment, clinical site, age, stroke type, side of hemiparesis and depression); Test type: Superiority or Other; p = 0.501, Regression, Logistic; Odds Ratio (OR) = 1.192, 95% CI 2-sided [0.715 to 1.985]

2. Primary Outcome: Walking Speed: Measured During a 10-meter Walk
Time Frame: Baseline and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
m/sec
  Baseline | 0.37 (0.22) | 0.38 (0.23) | 0.39 (0.22)
  12-month change from Baseline | 0.23 (0.20) | 0.24 (0.23) | 0.25 (0.22)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program; The second primary analysis assessed the timing effect and its interaction with initial severity of gait impairment on walking speed change from baseline to 1 year after stroke; Test type: Superiority or Other; p = 0.242, Regression, Linear — We did not formally conduct statistical inference on the timing effect because the first primary null hypotheses is accepted. The p-value provided is the smallest alpha level that one would claim significant difference between early- and late-LTP; Mean Difference (Final Values) = 0.01 — Even though there was no formal inference of timing effect, we still provided descriptive statistics for the 6-month and 12-month changes. In addition, paired t-tests were used to compare within-group improvements

3. Secondary Outcome: Percentage of Patients Who Successfully Improved Functional Level of Walking at 6 Months Post-stroke
Description: as for outcome 1
Time Frame: Baseline and 6 months post-stroke
Population: Intention to treat analysis. Missing data were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: percent of participants
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
percent of participants | 50.4 | 32.2 | 49.2
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program; Logistic regression was used to compare the proportion of participants who improved functional level of walking between early-LTP and Late-LTP (Usual Care) adjusting for pre-specified covariates (severity of impairment, clinical site, age, stroke type, side of hemiparesis and depression); Test type: Superiority or Other; p = 0.010, Regression, Logistic; Pairwise comparisons were conducted: Early-LTP versus Late-LTP, which had received only usual care in the 2- to 6-month post-stroke period; Odds Ratio (OR) = 1.94, 95% CI 2-sided [1.18 to 3.21]
Statistical Analysis 2: Comparison: Late Locomotor Training Program vs Home Exercise Program; Logistic regression was used to compare the proportion of participants who improved functional level of walking between HEP and Late-LTP (Usual Care) adjusting for pre-specified covariates (severity of impairment, clinical site, age, stroke type, side of hemiparesis and depression); Test type: Superiority or Other; p = 0.007, Regression, Logistic; Pairwise comparisons were conducted: HEP versus Late-LTP, which had received only usual care in the 2- to 6-month post-stroke period; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.22 to 3.42]

4. Secondary Outcome: 6 Month Outcome: Walking Speed: Measured During a 10-meter Walk
Time Frame: Baseline and 6 months post-stroke
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
m/sec
  Baseline | 0.37 (0.22) | 0.38 (0.23) | 0.39 (0.22)
  6 month change from Baseline | 0.25 (0.21) | 0.13 (0.14) | 0.23 (0.20)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program; 6 month secondary analysis. Following the overall ANOVA test, pairwise comparison was conducted to assess differences in walking speed changes between early-LTP and late-LTP; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Bonferroni adjustment for multiple testing was used in the pair-wise comparisons of the secondary outcomes. A difference is claimed to be statistically significant when p<0.0014; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.08 to 0.16]
Statistical Analysis 2: Comparison: Late Locomotor Training Program vs Home Exercise Program; 6 month secondary analysis. Following the overall ANOVA test, pairwise comparison was conducted to assess differences in walking speed changes between HEP and late-LTP; Test type: Superiority or Other; p < .0001, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [0.05 to 0.14]

5. Secondary Outcome: 6 Minute Walking Distance (Meters)
Description: Distance walked in 6 minutes.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
meters
  Baseline | 124.1 (77.5) | 125.7 (81.8) | 126.3 (75.0)
  6-month change from baseline | 81.8 (62.8) | 41.0 (47.4) | 75.9 (69.3)
  12-month change from baseline | 73.2 (69.4) | 79.0 (75.1) | 85.2 (72.9)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; Primary 12 month analysis. Paired t-tests were used to compare within-group improvements and ANOVA to assess differences across the three groups followed with pairwise comparisons; Test type: Superiority or Other; p = 0.45, ANOVA — Test differences across the three groups in change of 6 minute walking distance from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 6 month secondary analysis. Paired t-tests were used to compare within-group improvements and ANOVA to assess differences across the three groups followed with pairwise comparisons; Test type: Superiority or Other; p < 0.001, ANOVA; Test differences across the three groups in change of 6 minute walking distance from baseline to 6-month post stroke

6. Secondary Outcome: Step Activity Monitor (SAM)- Median of Average Number of Steps Per Day
Description: As measured with a step activity monitor averaged over 2 days.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Median (Inter-Quartile Range); unit: steps
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
steps
  Baseline | 1468 [601 to 3889] | 1664 [647 to 3354] | 1882.5 [905 to 3384]
  6-month change from Baseline | 1017 [-102 to 2209] | 565.5 [-362 to 2043] | 1357 [84 to 3382]
  12-month change from Baseline | 858 [-253 to 2422] | 1022 [-111 to 3009] | 1471 [435 to 3481]
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 12 month primary outcome. The Kruskal-Wallis procedure was used to assess differences across the three groups in number of steps taken in the community. Wilcoxon signed rank tests were used to compare within-group improvements; Test type: Superiority or Other; p = 0.10, Kruskal-Wallis; Test differences across the three groups in change of number of steps from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 6 month secondary analysis. The Kruskal-Wallis procedure was used to assess differences across the three groups in number of steps taken in the community. Wilcoxon signed rank tests were used to compare within-group improvements; Test type: Superiority or Other; p = 0.04, Kruskal-Wallis; Test differences across the three groups in change of number of steps from baseline to 6-month post stroke

7. Secondary Outcome: Stroke Impact Scale (SIS) - Participation
Description: Range = 0 - 100. The Stroke Impact Scale is a measure of function (including ADL-IADL and mobility) and quality of life (participation). The Participation Scale is a single domain of the Stroke Impact Scale in which participation is defined as the ability to engage in meaningful activities with 0 indicating inability to engage in any meaningful activities and 100 indicating the ability to fully engage in meaningful activities.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 45.0 (23.3) | 46.6 (23.0) | 44.8 (23.5)
  6 month change from Baseline | 11.8 (26.8) | 7.7 (20.5) | 14.7 (22.9)
  12 month change from Baseline | 17.1 (25.9) | 13.1 (22.0) | 14.4 (20.6)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 12 month primary outcome. Paired t-tests were used to compare within-group improvements and ANOVA to assess differences across the three groups followed with pairwise comparisons; Test type: Superiority or Other; p = 0.48, ANOVA; Test differences across the three groups in change of SIS Participation from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 6 month secondary outcome. Paired t-tests were used to compare within-group improvements and ANOVA to assess differences across the three groups followed with pairwise comparisons; Test type: Superiority or Other; p = 0.06, ANOVA; Test differences across the three groups in change of SIS Participation from baseline to 6-month post stroke

8. Secondary Outcome: Stroke Impact Scale (SIS) - Activities of Daily Living/Instrumental Activities of Daily Living (ADL/IADL)
Description: Range 0 - 100 The Stroke Impact Scale (SIS) is a measure of function including ADL/IADL. The ADL/IADL scale is a single domain of the Stroke Impact Scale in which ADL is defined as the ability to take care of basic needs and IADL is defined as the ability to perform activities that make it possible to live independently in the community, with 0 indicating complete dependence on others and 100 indicating the ability to live independently without difficulty.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 54.1 (20.1) | 55.7 (20.4) | 54.4 (20.7)
  6-month change from baseline | 9.8 (17.2) | 7.0 (17.8) | 13.0 (16.9)
  12-month change from baseline | 9.6 (19.5) | 9.4 (17.2) | 14.5 (19.0)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.07, ANOVA; Test differences across the three groups in change of SIS ADL/iADL from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.03, ANOVA; Test differences across the three groups in change of SIS ADL/iADL from baseline to 6-month post stroke

9. Secondary Outcome: Stroke Impact Scale (SIS) - Mobility
Description: Range = 0 - 100. The Stroke Impact Scale (SIS) is a measure of function including Mobility. The Mobility scale is a single domain of the Stroke Impact Scale which captures the ability to balance and move, with 0 indicating severe restrictions in balance and mobility and 100 indicating independence in mobility and balance.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 57.0 (22.1) | 60.5 (20.7) | 59.1 (19.5)
  6-month change from baseline | 15.3 (21.4) | 7.0 (15.7) | 14.9 (20.0)
  12-month change from baseline | 13.7 (21.6) | 12.0 (19.1) | 14.2 (20.3)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.69, ANOVA; Test differences across the three groups in change of SIS Mobility from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < .0001, ANOVA; Test differences across the three groups in change of SIS Mobility from baseline to 6-month post stroke

10. Secondary Outcome: Fugl-Meyer Lower Extremity Score
Description: Range 0 - 34 The Fugl-Meyer Lower Extremity Score measures your ability to move the lower extremity with 0 indicating no movement and 34 indicating the ability to selectively move the lower extremity without difficulty.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 23.7 (6.7) | 24.8 (6.4) | 24.7 (6.3)
  6-month change from Baseline | 2.2 (3.4) | 1.3 (3.3) | 2.4 (4.1)
  12-month change from Baseline | 1.7 (3.9) | 1.5 (3.7) | 2.5 (4.3)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; 12 month primary analysis. Paired t-tests were used to compare within-group improvements and ANOVA to assess differences across the three groups followed with pairwise comparisons; Test type: Superiority or Other; p = 0.13, ANOVA; Test differences across the three groups in change of FM-LE from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.04, ANOVA; Test differences across the three groups in change of FM-LE from baseline to 6-month post stroke

11. Secondary Outcome: Berg Balance Score
Description: Range = 0 - 56 The Berg Balance Score assesses balance in sitting, standing, reaching, shifting weight and turning, with 0 defined as inability to balance and 56 defined as the ability to balance independently and without difficulty while performing each task.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 35.0 (14.4) | 35.9 (14.1) | 36.5 (13.6)
  6-month change from Baseline | 8.8 (8.1) | 5.3 (7.0) | 7.9 (8.5)
  12-month change from Baseline | 8.0 (7.8) | 5.9 (9.1) | 8.3 (8.8)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.06, ANOVA; Test differences across the three groups in change of Berg Balance Score from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.001, ANOVA; Test differences across the three groups in change of Berg Balance Score from baseline to 6-month post stroke

12. Secondary Outcome: Activities Specific Balance Confidence (ABC) Score
Description: Range = 0 - 100 The ABC scale is a self reported measure of confidence with activities such as walking around the house, standing on a chair to reach or getting out of a car without losing balance or becoming unsteady. A score of 0 indicates no confidence that the activities can be performed without losing balance and a score 100 indicates confidence that the activities can be accomplished without losing balance.
Time Frame: Baseline, 6 months and 12 months post-stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Number analyzed (Participants) | 139 | 143 | 126
units on a scale
  Baseline | 43.6 (23.5) | 47.0 (25.4) | 44.5 (22.6)
  6-month change from Baseline | 13.8 (20.8) | 6.2 (20.2) | 15.6 (19.4)
  12-month change from Baseline | 11.2 (22.3) | 11.7 (22.1) | 13.9 (21.7)
Statistical Analysis 1: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.62, ANOVA; Test differences across the three groups in change of ABC score from baseline to 12-month post stroke
Statistical Analysis 2: Comparison: Early Locomotor Training Program vs Late Locomotor Training Program vs Home Exercise Program; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; Test differences across the three groups in change of ABC score from baseline to 6-month post stroke

ADVERSE EVENTS:
Time Frame: Total of 10 months from point of randomization at 2 months to the 12 month final assessment.
Description: Vital signs including heart rate, blood pressure and oxygen saturation were monitored every 5 minutes during exercise interventions. In addition monthly phone calls were used to capture rehospitalizations, recurrent stroke, MI, etc.
Arm/Group | Early Locomotor Training Program | Late Locomotor Training Program | Home Exercise Program
Serious Adverse Events (participants affected / at risk) | 51/139 | 59/143 | 39/126
Other Adverse Events (participants affected / at risk) | 100/139 | 101/143 | 88/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Locomotor Training Program (N=139) | Late Locomotor Training Program (N=143) | Home Exercise Program (N=126)
Recurrent Stroke (Vascular disorders) | 6 (6) | 3 (3) | 1 (1)
Myocardial Infarction (MI) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (8) | 5 (7)
Hospitalization (General disorders) | 45 (64) | 53 (83) | 31 (48)
Limitation in activities of daily living (ADL)>48hrs (General disorders) | 1 (1) | 2 (2) | 4 (4)
Other (General disorders) | 1 (1) | 1 (1) | 4 (4)
Death (General disorders) | 3 (3) | 4 (4) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Locomotor Training Program (N=139) | Late Locomotor Training Program (N=143) | Home Exercise Program (N=126)
Minor fall, no or minimal injury (General disorders) | 76 (181) | 77 (160) | 75 (150)
Open sore or blister, cuts (Skin and subcutaneous tissue disorders) | 8 (9) | 9 (10) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle soreness or pain that persists for more than 48 hours (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (12) | 10 (10)
Dizziness/Fainting (General disorders) | 11 (11) | 8 (9) | 0 (0)
Diaphoretic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0)
Excessive hypertension during exercise that requires the intervention to be stopped for the day (Cardiac disorders) | 5 (6) | 8 (8) | 10 (11)
Low blood pressure during exercise that requires intervention to be stopped for the day (Cardiac disorders) | 8 (11) | 7 (7) | 2 (3)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Other (General disorders) | 42 (59) | 47 (89) | 28 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No